CLINICAL TRIAL: NCT03432754
Title: Health Education and Lifestyle Training in Older Adults
Acronym: HEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ruchika Prakash, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014B0337
Record Dates: First submitted 2018-02-07; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Older Adults
Keywords: Older adults; Mindfulness; Mind wandering; Health education; Working memory; Cognitive functioning; Emotion regulation; Emotional functioning
MeSH Terms: conditions — Health Education; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This randomized control trial compared a mindfulness-based attention training (MBAT) group with an active control lifestyle education group. A total of 147 individuals underwent eligibility screening over the phone and in-person at an initial assessment session. Of those eligible, 75 participants volunteered to participate and were randomly assigned to groups. However, one of these participants did not complete the first assessment session and was randomized in error. Thus, 74 participants who completed the first assessment session and met all eligibility criteria were randomly assigned to either the MBAT group or the active control group (lifestyle education). Randomization was conducted by a study author using a computerized random number generator program (randomization.com), applying a varying block size of two and four and stratifying participants by gender. A total of 37 participants were allocated to the each of the two groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization was conducted by the principle investigator (PI) and study coordinator using a computerized random number generator program (randomization.com). All experimenters (except the PI and study coordinator) were blinded to group assignments until study conclusion. To further reduce demand characteristics, participants were unaware of which group was considered the experimental intervention until debriefed by an experimenter after completing the study. Study binders were created to blind group assignment, and participants in each group were asked not to discuss the sessions with members of the other group or with the experimenter at their post-intervention assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Attention Training (Experimental): Four weekly group mindfulness attention training sessions of a 1.5-hour duration. Participants provided with audio recordings, readings, and homework assignments consisting of various mindfulness practices.
  Interventions: Behavioral: Mindfulness-Based Attention Training
- Lifestyle Education Group (Active Comparator): Four weekly group lifestyle education sessions of a 1.5-hour duration. Homework consisting of reading, diet monitoring, stretching/toning exercises, and brainstorming new healthy living techniques/ideas.
  Interventions: Behavioral: Lifestyle Education

INTERVENTIONS:
Behavioral: Mindfulness-Based Attention Training — The mindfulness-based attention training is closely modeled after the traditional mindfulness-based stress reduction (MBSR) protocol, it incorporates formal MBSR practices such as breath exercises, body scans and long sitting meditations. Specifically, MBAT is an abbreviated version of MBSR with a focus on the cognitive components.
  Arms: Mindfulness-Based Attention Training
Behavioral: Lifestyle Education — The control group, which will be used to compare the effects of mindfulness training on emotional and cognitive functioning and mind wandering in older adults, will comprise of scientific health and lifestyle information. Lectures will be focused on concepts presented in the book "The Culprit and the Cure: Why lifestyle is the culprit behind America's poor health and how transforming that lifestyle can be the cure." Meetings will cover how to begin and maintain a more nutritious diet, classifying healthy choices across food groups, completing stretching/toning exercises, and reviewing homework.
  Arms: Lifestyle Education Group

SUMMARY:
The investigators conducted a mindfulness training intervention in older adults aimed at examining the effects of brief mindfulness training on mind wandering as well as the cognitive and affective functioning of older adults. Individuals completed pre- and post-assessments of mind wandering and cognitive functioning. Additionally, all participants completed neuropsychological measures and self-report questionnaires.

DETAILED DESCRIPTION:
Age-related differences in sustained attention may be related to the prevalence and content of task unrelated thought or mind-wandering. Older adults report less mind-wandering in sustained tasks than younger adults, something that is surprising due to the reduced performance on tasks. It is clear that both cognitive and emotional processes underlie comprehension and sustained attention and relate to prevalence of task unrelated thought and performance. A complex process such as reading comprehension presents a challenge for improvement because of the wide range of changes that occur with age. Pharmacological therapies can target only a limited number of the many changes believed to underlie functional decline. One way that may mitigate these declines in performance in a broad way is mindfulness training. Thus, the investigators conducted a randomized study to assess the effects of mindfulness training relative to an active health education control group on mind wandering and controlled processing abilities in older adults. All individuals that contact the Clinical Neuroscience Laboratory (CNLab) with interest underwent a phone screening assessing inclusion/exclusion criteria.Those participants meeting I/E criteria were invited to participate in the study. During the first assessment session, written informed consent was obtained; additional inclusion/exclusion measures were administered; and self-report questionnaires and assessment measures were completed. Following the first assessment session, four training sessions took place. Participants were randomized into either the a mindfulness training intervention or a health education intervention. Subsequently, all participants were invited back for post-assessment session.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 74 years of age
* No prior exposure to mindfulness training
* No significant meditation experience
* Have never engaged in regular practices of yoga
* Capable of attending both assessment and training sessions
* Corrected (near and far) visual acuity of 20/40 or better
* Normal color vision
* No self-reported history of psychiatric, neurological, or chronic inflammatory conditions
* Absence of psychiatric medication use
* Native English Speaker
* Adequate performance on the Mini-Mental Status Examination (MMSE; >23)
* Depression score on the Geriatric Depression Scale (GDS) below clinical level (<10)

Exclusion Criteria:

* Below 60 years of age or above 74 years of age
* Have exposure to or experience with any type of meditation or yoga regularly (one hour a week for at least 12 months)
* Any physical or pragmatic limitation that prohibits attendance at both sessions
* Corrected (near or far) visual acuity worse than 20/40
* All types of color blindness
* Presence of diagnosed neurological disorders (such as: Alzheimer's disease, Parkinson's disease or multiple sclerosis) or chronic inflammatory conditions
* Presence of any diagnosed psychiatric disorder such as depression, attention deficit hyperactivity disorder (ADHD), substance abuse
* Presence of psychiatric medication use such as Xanax, Wellbutrin, or Vivance
* Non-Native English Speaker or no fluency in English
* Inadequate performance on the Mini-Mental Status Examination (MMSE; <23)
* Depression score on GDS indicative of clinical depression (>10)

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2015-04-29 (Actual); Study Completion 2015-04-29 (Actual)

PRIMARY OUTCOMES:
Change in Global Performance on Computerized Attentional Control Tasks | Baseline and after the 4-week intervention
  Signal detection scores on two computerized tasks of attentional control calculated for each task using the formula for logistic distributions: dL = ln{[H(1-FA)]/[(1-H)FA]}, where H refers to hit rates and FA refers to false alarms.
Change in Mind-Wandering During Attentional Control Tasks | Baseline and after the 4-week intervention
  Frequency with which thoughts categorized as evaluating performance or off-task in response to quasi-random mind-wandering probes collected during two computerized tasks of attentional control.

SECONDARY OUTCOMES:
Change in Self-report Mindful Attention Awareness Scale (MAAS) | Baseline and after the 4-week intervention
  Self-reported current level of dispositional mindfulness assessed using 15-item Mindful Attention Awareness Scale (MAAS). Each item is scored from 1-6 and then averaged to get a total score between 1-6 with higher scores reflecting higher levels of dispositional mindfulness.
Change on Self-Report Measure of Emotion Dysregulation | Baseline and after the 4-week intervention
  Changes in emotion dysregulation assessed using the 36-item Difficulties in Emotion Regulation Scale (DERS). Each items is scored 1-5 with a total score between 36-180 with a higher score reflecting greater emotion dysregulation.
Change in Local Metrics of Attentional Control During Go/No-Go Task | Baseline and after the 4-week intervention
  Changes in reaction time and accuracy preceding mind-wandering probes during one of the attentional control tasks, the Go/No-Go Task.

CONTACTS AND LOCATIONS:
Overall Officials: Ruchika Prakash, PhD, Principal Investigator — Ohio State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fountain-Zaragoza S, Londeree A, Whitmoyer P, Prakash RS. Dispositional mindfulness and the wandering mind: Implications for attentional control in older adults. Conscious Cogn. 2016 Aug;44:193-204. doi: 10.1016/j.concog.2016.08.003. Epub 2016 Aug 16. PMID 27541935
- [Derived] Duraney EJ, Phansikar M, Prakash RS. Psychosocial Correlates of Adherence to Mind-Body Interventions. Prev Sci. 2025 Jul;26(5):839-848. doi: 10.1007/s11121-025-01810-1. Epub 2025 May 6. PMID 40325320